CLINICAL TRIAL: NCT06252311
Title: The Effect of Mindfulness-Based Breastfeeding Programme on Breastfeeding Awareness and Breastfeeding Attitude in Mothers After Cesarean Delivery: A Randomised Controlled Study
Brief Title: The Effect of Mindfulness-Based Breastfeeding Programme in Mothers After Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Serife BUYUKOKUDAN, Sub-Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AkdenizU-HF-SB-01
Record Dates: First submitted 2024-02-02; First posted 2024-02-09 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-05

CONDITIONS: Breastfeeding
Keywords: Mindfulness; Breast Feeding; Attitude; Nursing
MeSH Terms: conditions — Breast Feeding; Behavior

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups with a Mindfulness-Based Breastfeeding Programme and control group
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, the researcher will not be blinded during the intervention implementation and data collection via telephone interviews. However, the control group will receive general breastfeeding education, allowing for participant blinding. Randomisation will be performed by an independent statistician using randomly generated numbers. Additionally, blinding of statisticians will be implemented during data entry and analysis by labelling primiparas in the experimental group as Xa and multiparas as Xb, and primiparas in the control group as Ya and multiparas as Yb
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Breastfeeding Programme group (Experimental): Participants in the experimental group will receive the Mindfulness-Based Breastfeeding Programme, which consists of six 30-minute sessions within 0-72 hours. They will also be asked to complete a personal information form. In addition to the hospital sessions, educational materials, including home applications and audio recordings, will be sent via WhatsApp after discharge. During the first week after discharge, counselling will be provided by phone on the continuation of mindfulness-based practices, continuation of breastfeeding and problems related to breastfeeding, and referral to the health facility in case of problems, "Iowa Infant Feeding Attitude Scale" and "Mindful Breastfeeding Scale" will be administered by phone call in the 2nd month and finally the "Infant Feeding Follow-up Form" prepared by the researcher based on the literature will be used to assess the continuity of breastfeeding in the 1st week, 2nd month, 4th month and 6th month.
  Interventions: Behavioral: Mindfulness-Based Breastfeeding Programme
- Control group (No Intervention): After the women in the control group have been informed about the study and have given their consent, they will complete a personal information form and then they will receive routine breastfeeding support and standard hospital care. The control group will be administered the Iowa Infant Feeding Attitude Scale and the Mindful Breastfeeding Scale by telephone interview at month 2 and the Infant Feeding Follow-up Form at week 1, month 2, month 4 and month 6.

INTERVENTIONS:
Behavioral: Mindfulness-Based Breastfeeding Programme — Mindfulness-Based Breastfeeding Programme will consist of structure and anatomy of the breast and milk production, breast milk content, benefits of breast milk, breast care, frequency and duration of breastfeeding, correct and comfortable position for breastfeeding, effects of stress on lactation hormones and milk production, World Health Organization guidelines on duration and continuity of breastfeeding, time to start complementary feeding general information on recommendations, General information about breastfeeding with awareness, mentioning its purpose and programme flow, and it includes formal and informal practices such as breathing awareness exercises, noticing the autopilot, lying/sitting meditation, body scanning exercises and mindful breastfeeding practice.
  Arms: Mindfulness-Based Breastfeeding Programme group

SUMMARY:
The study is a randomised controlled trial designed to determine the effect of the Mindfulness-Based Breastfeeding Programme on maternal breastfeeding awareness, breastfeeding attitudes and breastfeeding continuation among mothers who have given birth by caesarean section. The study will evaluate the effectiveness of the Mindfulness-Based Breastfeeding programme using the "Mindful Breastfeeding Scale" and "Iowa Infant Feeding Attitude Scale". The research will use stratified and simple randomisation methods. Research data will be collected from mothers who gave birth by caesarean section at the gynaecology clinic of the Afyonkarahisar Health Sciences University Health Application and Research Center of between April 2024 and December 2025.

DETAILED DESCRIPTION:
Breastfeeding is an ideal form of nutrition that has important implications for the health of mothers, infants and society. In addition to its beneficial effects on biopsychosocial health, it also contributes to social development in economic terms. Because of the powerful effects of breastfeeding, various studies, practices and guidelines have been organised for the initiation and maintenance of breastfeeding. World Health Organization recommends initiation of breastfeeding within the first hour after birth, exclusive breastfeeding for the first 6 months and continued breastfeeding with complementary foods until the age of 2 years. However, in Turkey, exclusive breastfeeding for the first 6 months is 41% and the median duration of breastfeeding is 16.7 months. Although most women are willing and able to breastfeed, there are several factors that affect the initiation and continuation of breastfeeding. Studies of the difficulties in initiating and maintaining breastfeeding may portray breastfeeding as primarily a challenging and demanding behaviour, rather than a reciprocal act that provides a positive emotional exchange for both infant and mother. Mindfulness-based breastfeeding involves focusing on the present moment and experiencing breastfeeding moment by moment. This approach is based on the idea that breastfeeding is a time for the mother and baby to relax and is a natural process. It is believed that mindfulness-based breastfeeding can have positive effects. While there are studies in the international literature on the effects of mindfulness practices during pregnancy on breastfeeding, mindfulness-based childbirth education interventions, transition to mindfulness-based motherhood, and the effects of mindfulness-based practices on maternal self-efficacy, no study has evaluated the effect of a mindfulness-based breastfeeding programme on breastfeeding attitude and awareness after a cesarean section. This randomised controlled study was planned to investigate the effect of a mindfulness-based structured breastfeeding programme on breastfeeding awareness and breastfeeding attitude after caesarean section. In order to determine the sample size, 70 experimental and 70 control groups were determined to be sufficient according to the power analysis performed by using the G*Power programme version 3.1 when the type-I error level (α)=0.05 and the power of the study was accepted as 0.90. Considering that women could not be provided with appropriate training due to pain and anaesthesia effect after caesarean section, sessions lasting 30 minutes were planned at hours when they felt comfortable and ready within 0-72 hours. The women in the experimental group will be trained a total of 6 sessions of mindfulness-based breastfeeding programme will be implemented, while the control group will be given rutin care. The research data will be collected by using Personal Information Form including sociodemographic characteristics, Iowa Infant Feeding Attitude Scale, Mindful Breastfeeding Scale and Infant Feeding Follow-up Form. As a result of the study, it is expected that breastfeeding awareness, breastfeeding attitude scores and breastfeeding continuity of the experimental group will be higher than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40
* Having had a caesarean section at 37 weeks or more of gestation
* Having been hospitalised at Afyonkarahisar Health Sciences University Health Application and Research Center, Gynaecology and Obstetrics Clinic
* Having a single and healthy baby (no multiple pregnancy)
* Having completed at least primary school
* Being able to communicate in Turkish by phone using the WhatsApp application
* The baby is with the mother

Exclusion Criteria:

* Having a high-risk pregnancy
* Having a medical condition or taking medication that prevents breastfeeding
* Having a communication problems (vision, hearing, speech, language problems)
* Having a psychiatric illness
* Hysterectomy after caesarean section
* There is an obstacle that prevents the baby from being with the mother or being in the neonatal intensive care unit
* Having a condition/disease that prevents you from doing mindfulness practices (breathing exercises, body scanning)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Mindful Breastfeeding Scale (MIND-BFS) | In the 2nd month after implementing the mindfulness-based breastfeeding program
  Evaluation of the effect of mindfulness-based breastfeeding programme on postpartum breastfeeding awareness in women who underwent cesarean section.
  The Mindful Breastfeeding Scale (MIND-BFS), is a 9-item instrument that assesses mindfulness-based breastfeeding practice in the postpartum period. The scale is unidimensional and developed in 5-point Likert format. The answers to the scale items vary from (1) always (5) never. The total score obtained from the scale ranges from 9 to 45, and as the total score obtained from the scale increases, the level of breastfeeding awareness increases. The Cronbach's alpha value of the scale was found to be 0.83.
Iowa Infant Feeding Attitude Scale (IIFAS) | In the 2nd month after implementing the mindfulness-based breastfeeding program
  Evaluation of the effect of mindfulness-based breastfeeding programme on postpartum breastfeeding attitude in women who underwent caesarean section.
  The Iowa Infant Feeding Attitude Scale (IIFAS) was to assess women's attitudes towards breastfeeding and predict the duration of breastfeeding and choice of infant feeding method. The scale comprises 17 items, each rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The scale includes 9 positive items about breastfeeding and 8 positive items about formula feeding, with the latter being reverse scored (1=5, 2=4, 4=2 and 5=1). The total attitude score ranges from 17 points (indicating a positive attitude towards bottle feeding) to 85 points (indicating a positive attitude towards breastfeeding).

SECONDARY OUTCOMES:
Infant Follow-up Form | 1st week, 2nd month, 4th month and 6th month after birth
  Evaluation of the effect of mindfulness-based breastfeeding programme on the continuity of breastfeeding in women who underwent caesarean section. This is a 7-question form designed by the researcher to assess the continuity of breastfeeding at specific time intervals, including questions such as adequate weight gain of the baby, breastfeeding status and feeding method

CONTACTS AND LOCATIONS:
Overall Officials: Oznur KORUKCU, Principal Investigator — Akdeniz University
Locations (2):
- Turkey (Türkiye) (2):
  - Afyonkarahisar Health Sciences University Health Application and Research Center, Afyonkarahisar, Dörtyol
  - AFSU Health Research and Application Center, Afyonkarahisar, Merkez

IPD SHARING:
Plan to Share IPD: No